CLINICAL TRIAL: NCT01173523
Title: A Phase II Study of the Hsp90 Inhibitor, STA-9090, in Patients With Relapsed or Refractory Small Cell Lung Cancer
Brief Title: Study of Hsp90 Inhibitor, STA-9090 for Relapsed or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David M. Jackman, MD (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor-Investigator, David M. Jackman, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-048
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Small Cell Lung Cancer
Keywords: Hsp90 Inhibitor; relapsed; refractory
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: STA-9090 (Experimental): Once weekly IV dosing of STA-9090 200mg/m2 was given weeks 1, 2, and 3 of a 4-week cycle. Participants received treatment until evidence of progressive disease or unacceptable toxicity. Participants were stratified at baseline into 2 distinct prognostic groups. Cohort A participants had relapsed > 60 days following initial chemotherapy completion.
  Interventions: Drug: STA-9090
- Cohort B: STA-9090 (Experimental): Once weekly IV dosing of STA-9090 200mg/m2 was given weeks 1, 2, and 3 of a 4-week cycle. Participants received treatment until evidence of progressive disease or unacceptable toxicity. Participants were stratified at baseline into 2 distinct prognostic groups. Cohort B participants had not responded or had relapsed </= 60 days from the completion of initial chemotherapy.
  Interventions: Drug: STA-9090

INTERVENTIONS:
Drug: STA-9090
  Other Names: Ganetespib

SUMMARY:
Small cell lung cancer (SCLC) is a chemotherapy and radiotherapy sensitive tumor, but with very high rates of relapse and metastasis, resulting in a very poor outcome. Among limited-stage patients, the relapse rate is at least 80% and among extensive-stage patients, the relapse rate is 95-98%. The impetus to develop more effective therapies against novel targets in SCLC is therefore high.

Hsp-90 inhibitors are a new class of drugs with important anti-malignant potential in a variety of tumor types because of the reliance of multiple oncoproteins on Hsp90 function. Although small cell neuroendocrine tumors generally carry many mutated oncoproteins, without clearly defined clients for Hsp90 mediating inhibitor effects in these cells, a recent study demonstrated that Hsp90 inhibition causes massive apoptosis by activating the intrinsic apoptotic pathway in a number of SCLC cell lines. SCLC is a particularly attractive target for apoptosis inducing drugs because of high growth rates and evidence of molecular alterations affecting apoptotic mechanisms.

STA-9090 is a novel, small-molecule inhibitor of Hsp90. Unlike earlier generations of Hsp90 inhibitors, STA-9090 has been shown to be a potent inducer of apoptosis in a variety of cell lines and has anti-tumor activity in multiple types of human xenografts. As was seen with other Hsp90 inhibitors, STA-9090 also induces apoptosis in a number of SCLC cell lines.

Based on the anti-tumor potential seen pre-clinically with Hsp90 inhibition, the potent effects of STA-9090 seen pre-clinically as compared with other inhibitors in the same class, as well as early data suggesting safety and tolerability of this drug in the Phase I setting, we propose to study the single-agent activity of STA-9090 in a Phase II trial of patients with relapsed or refractory small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective

* To determine the progression-free rate at 8 weeks in participants with relapsed or refractory small cell lung cancer who have received <3 prior regimens of systemic chemotherapy

Secondary Objectives

* To determine the response rate using radiologic assessment according to standard RECIST 1.1 criteria
* To determine median progression free survival and overall survival
* To characterize the toxicity profile of STA-9090 in this patient population

Exploratory Objectives

* To analyze levels of circulating tumor cells (CTCs) from blood samples obtained serially throughout the study and assess the utility of measuring these cell subsets as a marker of disease burden as well as response to therapy
* To analyze the participant population by identification of gene expression profiles (measured in RNA from available tumor biopsies) associated with the efficacy and resistance to STA-9090

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of small cell lung cancer and confirmed progressive disease by radiographic study
* </= 3 prior chemotherapy regimens
* Subjects with brain metastases will be allowed if they have been treated with surgery and/or radiation therapy > 21 days prior, are asymptomatic, and are stable for at least 1 week off steroids
* Must have measurable disease
* >/= 18 years of age
* Life expectancy of greater than 12 weeks
* EGOG performance status 0 or 1
* Lab values must be within limits outlined in the protocol
* Not pregnant or breastfeeding
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Chemotherapy or radiotherapy within 3 weeks or within 5 half-lives of previous therapy
* History of severe allergic or hypersensitivity reactions to taxanes.
* Subjects who have not recovered from adverse events or toxicities due to agents administered more than 4 weeks earlier to a grade 1 or less
* Not receiving any other study agents
* History of or current coronary artery disease, myocardial infarction, angina pectoris, angioplasty or coronary bypass surgery.
* Baseline QTc > 470 msec or previous history of QT prolongation while taking other medications.
* Ventricular ejection fraction of < 55%.
* History or current uncontrolled dysrhythmias, or requirement for antiarrhythmic medications, or Grade 2 or greater left bundle branch block.
* ECG with clinically significant ventricular arrhythmias or ischemia
* Major surgery within 4 weeks of starting treatment
* Poor venous access necessitating use of indwelling catheter for IV therapy
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance
* History of another malignancy unless disease-free for 3 years and deemed to be at low risk for recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07-28 (Actual); Primary Completion 2013-06-07 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jackman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massacusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from July 2010 through March 2013.
Period: Overall Study
Arm/Group | Cohort A: STA-9090 | Cohort B: STA-9090
Started | 13 | 12
Completed | 0 (Since treatment was not of fixed duration, all participants were considered as 'Not Completed'.) | 0 (Since treatment was not of fixed duration, all participants were considered as 'Not Completed'.)
Not Completed | 13 | 12
Not completed — Clinical Progression | 1 | 1
Not completed — Progressive Disease | 10 | 8
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: STA-9090 | Cohort B: STA-9090 | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 72] | 59.5 [43 to 70] | 61 [43 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: 8-Week Progression-Free Rate
Description: The 8-week progression free rate is defined as the percentage of participants achieving complete response (CR), partial response (PR) or stable disease (SD) based on RECIST 1.1 criteria by the time of the first disease assessment (8 weeks). Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions; PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD; and SD is neither sufficient decrease to qualify as PR nor sufficient increase to qualify as progressive disease (PD). PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. Response needed confirmation within 4 weeks. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: Disease was evaluated radiographically at baseline and every 8 weeks on treatment; Treatment continued until disease progression or unacceptable toxicity. Relevant for this endpoint was the first 8 week disease re-assessment.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: STA-9090 | Cohort B: STA-9090
Number analyzed (Participants) | 13 | 12
percentage of participants | 0.0 [0.0 to 24.7] | 8.3 [0.2 to 38.5]

2. Secondary Outcome: Overall Response Rate
Description: The objective response rate (ORR) was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiographically at baseline and every 8 weeks on treatment. Treatment duration was a median of 2 cycles (parallel to 2 months given the 4 week cycle length) and range of 1-2 cycles in this study cohort.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: STA-9090 | Cohort B: STA-9090
Number analyzed (Participants) | 13 | 12
percentage of participants | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 26.5]

3. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) based on the Kaplan-Meier method is defined as the time from study entry to the earliest documentation of disease progression (PD) based on RECIST 1.1 criteria or death. Participants alive without evidence of PD were censored at the date of last adequate disease assessment. Per RECIST 1.1 for target lesions PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression is appearance of one or more new lesions and/or unequivocal progression on existing non-target lesions.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: STA-9090 | Cohort B: STA-9090
Number analyzed (Participants) | 13 | 12
months | 1.61 [1.61 to NA] — Follow-up is not long enough/Data is not mature to provide upper bound 95% CI. | 1.81 [1.15 to NA] — Follow-up is not long enough/Data is not mature to provide upper bound 95% CI.

4. Secondary Outcome: Overall Survival
Description: Overall survival estimated using Kaplan-Meier (KM) methods is defined as the time from study entry to death due to any cause or date last known alive.
Time Frame: Long-term follow-up for survival occurred every 4 weeks. As of this analysis, follow-up among survivors was a median (range) of 11.5 months (0.9-47.9).
Population: The analysis dataset is comprised of treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: STA-9090 | Cohort B: STA-9090
Number analyzed (Participants) | 13 | 12
months | 4.96 [3.45 to NA] — Follow-up is not long enough/Data is not mature to provide upper bound 95% CI. | 6.70 [2.27 to NA] — Follow-up is not long enough/Data is not mature to provide upper bound 95% CI.

ADVERSE EVENTS:
Time Frame: Assessed weekly on treatment from time of first dose and up to day 30 post-treatment. Treatment duration was a median of 2 cycles (parallel to 2 months given the 4 week cycle length) and range of 1-2 cycles.
Description: Maximum grade toxicity by type for a patient over time including only events with treatment-attribution of possibly, probably or definitely was first calculated. Serious and Other AEs were defined as events of grades 3-5 and grades 1-2, respectively, based on CTCAEv3 which includes coding events as 'Other'. A patient appears only once for a given type of toxicity. Patients with reports of multiple toxicities of different types are reported multiple times under the relevant toxicity categories.
Arm/Group | Cohort A: STA-9090 | Cohort B: STA-9090
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 4/13 | 3/12
Other Adverse Events (participants affected / at risk) | 7/13 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: STA-9090 (N=13) | Cohort B: STA-9090 (N=12)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1
Allergic reaction (Immune system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Chills (General disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eye disorders - Other (Eye disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Flushing (Vascular disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 1
Infusion related reaction (General disorders) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Serum amylase increased (Investigations) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Weight loss (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: STA-9090 (N=13) | Cohort B: STA-9090 (N=12)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Alkaline phosphatase increased (Investigations) | 1 | 1
Allergic reaction (Immune system disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2
Chills (General disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 7
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eye disorders - Other (Eye disorders) | 1 | 0
Fatigue (General disorders) | 2 | 3
Flushing (Vascular disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2
Infections and infestations - Other (Infections and infestations) | 1 | 0
Infusion related reaction (General disorders) | 0 | 1
Lipase increased (Investigations) | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Serum amylase increased (Investigations) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Weight loss (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No